CLINICAL TRIAL: NCT06990542
Title: RAdiation Dose TAiloRing Guided by Enhanced Targeting
Brief Title: Image-guided, Tumor-focused Radiotherapy Treatment in Intermediate and High-risk Prostate Cancer
Acronym: RAD-TARGET
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University of California, San Diego (Other)
Responsible Party: Principal Investigator, Tyler Seibert, Radiation Oncologist, University of California, San Diego
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 812494
Record Dates: First submitted 2025-05-18; First posted 2025-05-25 (Actual); Last update posted 2025-06-29 (Actual); Status verified 2025-06

CONDITIONS: Prostate Cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care dose radiotherapy (No Intervention): Standard dose radiation therapy
- Tumor-focused radiotherapy (Experimental): Image-guided tumor-focused radiation therapy
  Interventions: Radiation: Image-guided tumor-focused radiation therapy

INTERVENTIONS:
Radiation: Image-guided tumor-focused radiation therapy — Image-guided tumor-focused radiation therapy
  Arms: Tumor-focused radiotherapy

SUMMARY:
This is a phase II non-blinded randomized controlled trial of image-guided, tumor-focused radiotherapy in patients with intermediate- or high-risk prostate cancer planning to undergo definitive radiotherapy with or without systemic therapy. The image-guided, tumor-focused radiotherapy will be compared to standard, whole-prostate treatment. The investigators hypothesize that tumor-focused radiotherapy reduces the radiation dose to organs close to the prostate, possibly leading to decreased acute toxicity to the genitourinary and gastrointestinal organs. The investigators will measure acute and late genitourinary and gastrointestinal toxicity due to radiation and regardless of cause. The investigators will also measure overall survival, metastasis-free survival, and quality of life, as well as biomarkers that may help predict, in the future, who may have a worse toxicity following radiation therapy.

DETAILED DESCRIPTION:
Definitive radiation therapy for prostate cancer with dose intensification and/or focal boosting has excellent oncologic outcomes. However, many patients experience long-term toxicity in particular to the genitourinary and gastrointestinal organs, impacting their quality of life. Given the excellent survivorship after definitive prostate cancer treatment, there is interest in identifying strategies that can improve the therapeutic ratio and minimize toxicity while maintaining excellent oncologic outcomes. Intraprostatic recurrence after definitive radiation therapy occurs at the site of the primary tumor and the dose to the site of the primary tumor is an important predictor of future treatment failure. This leads to the hypothesis that, if accurate discrimination between tumor(s) and benign prostate tissue can be achieved, radiation oncologists can devise tumor-focused radiation therapy plans that deliver ablative dose radiation therapy to the tumor(s) and de-escalated dose to the remainder of the electively irradiated prostate. This strategy is now possible thanks to advanced imaging technologies that can accurately identify the primary clinically significant tumor(s) to be targeted. De-escalated dose to the remainder of the prostate may lead to low dose also to neighboring organs, such as rectum and bladder, potentially leading to lower rates of acute and late toxicity and minimizing the impact of prostate cancer treatment on quality of life. A randomized trial is required to compare the efficacy and toxicity of tumor-focused radiation therapy to that of standard radiation therapy for definitive treatment of localized prostate cancer.

ELIGIBILITY:
Inclusion Criteria:

* Provision of signed and dated informed consent form
* Stated willingness to comply with all study procedures and availability for the duration of the study
* At least 18 years old
* Histologic confirmation of prostate adenocarcinoma with plan for curative-intent radiation therapy
* Lesion visible on prostate Magnetic Resonance Imaging and/or Prostate-Specific Membrane Antigen Positron Emission Tomography-Computed Tomography (according to the treating physician) with concordant pathology from biopsy needle locations.
* For participants able to cause a pregnancy: use of condoms or other methods to ensure effective contraception with partner during the radiation therapy treatment and for at least 6 months afterward.

Exclusion Criteria:

* Bilateral hip implants
* Prior prostatectomy
* Prior prostate cancer treatment (for example, focal therapy). Note that participants who started hormone therapy within the 90 days prior to randomization are eligible, as long as study-compatible imaging was performed within the 4 months prior to starting the hormone therapy.
* Prior radiation therapy to an area requiring treatment in the present study

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Prostate cancer
Enrollment: 150 (Estimated)
Dates: Start 2025-06-09 (Actual); Primary Completion 2028-12 (Estimated); Study Completion 2033-12 (Estimated)

PRIMARY OUTCOMES:
Acute toxicity | 3 months
  Acute any attribution genitourinary or gastrointestinal toxicity (grade 2 or higher), compared between randomized arms, defined as the percentage of patients with Common Terminology Criteria for Adverse Events genitourinary or gastrointestinal toxicity of grade 2 or higher within 3 months of completing radiation therapy.
  Based on the Common Terminology Criteria for Adverse Event, grade 1 is the lowest and grade 5 is the highest. Grade 5 represents the worst outcome (death).

CONTACTS AND LOCATIONS:
Overall Officials: Tyler Seibert, MD, PhD, Principal Investigator — University of California, San Diego
Locations (1):
- University of California, San Diego, La Jolla, California, United States

IPD SHARING:
Plan to Share IPD: No